CLINICAL TRIAL: NCT05947812
Title: A Clinical Evaluation of the Safety and Efficacy of Randomized Placebo Versus the 8-aminoquinoline Tafenoquine for Early Symptom Resolution in Patients With Mild to Moderate COVID 19 Disease and Low Risk of Disease Progression (the "ACLR8-LR" Study)
Brief Title: A Clinical Evaluation of the Safety and Efficacy of Randomized Placebo Versus the 8-aminoquinoline Tafenoquine for Early Symptom Resolution in Patients With Mild to Moderate COVID 19 Disease and Low Risk of Disease Progression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: 60P Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ 2022-08
Record Dates: First submitted 2023-07-13; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: COVID 19 Disease; Mild to Moderate COVID 19 Disease; SARS-CoV-2; Infectious Disease; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — Communicable Diseases | interventions — tafenoquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tafenoquine (Experimental): Tafenoquine two tablets 1x/day on Days 1, 2, 3, and then weekly (Days 10 ± 1 day, 17 ± 2 days, 24 ± 2 days, 31 ± 2 days and 38 ± 2 days) until sustained clinical recovery
  Interventions: Drug: Tafenoquine Oral Tablet
- Placebo (Placebo Comparator): Placebo two tablets 1x/day on Days 1, 2, 3, and then weekly (Days 10 ± 1 day, 17 ± 2 days, 24 ± 2 days, 31 ± 2 days and 38 ± 2 days) until sustained clinical recovery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tafenoquine Oral Tablet — Patients will be randomized and will receive and self-administer 200 mg Tafenoquine on Days 1, 2, 3, and then weekly (Days 10 ± 1 day, 17 ± 2 days, 24 ± 2 days, 31 ± 2 days and 38 ± 2 days) until sustained clinical recovery.
  Other Names: KODATEF™; Arakoda
  Arms: Tafenoquine
Drug: Placebo — Patients will be randomized and will receive and self-administer 200 mg Tafenoquine or matching placebo on Days 1, 2, 3, and then weekly (Days 10 ± 1 day, 17 ± 2 days, 24 ± 2 days, 31 ± 2 days and 38 ± 2 days) until sustained clinical recovery.
  Arms: Placebo

SUMMARY:
A clinical study to assess the efficacy and safety of oral tafenoquine compared to placebo in patients with mild to moderate COVID 19 disease and low risk of disease progression (the "ACLR8-LR" study).

DETAILED DESCRIPTION:
The TQ 2020_08 study is a double-blind placebo-controlled, Phase 2b clinical trial that plans to enroll approximately 148 non-hospitalized patients with mild to moderate COVID 19 disease and low risk of disease progression (the "ACLR8-LR" study). Patients will undergo a brief screening period before being randomized to receive either self-administered 200 mg tafenoquine or matching placebo for up to 38 days. Following the treatment period, patients will have a follow up visit at study Day 42. The study's primary efficacy endpoint is time to sustained clinical recovery from COVID-19 symptoms (4 uninterrupted days of aggregate symptom scores ≤ 2) through Day 28 (± 2 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18, regardless of COVID-19 vaccination status;
2. Laboratory confirmed infection COVID-19 disease as determined using an FDA-authorized COVID-19 rapid antigen test;
3. Able and willing to give written informed consent;
4. Willing to complete the following study activities and assessments:

   1. Keep an electronic diary from Study Days 2 through 42.
   2. Have phone or videoconferences with study team personnel on Study Days 10, 21, and 35.
   3. Have study samples collected in-home on Days 5, 14, 28, and 42
   4. Agree to return to clinic for additional safety evaluations if needed, as determined by the study team;
5. An aggregate patient-reported COVID-19 symptom score of at ≥3 on the first day of drug administration (Study Day 1).
6. Must agree not to enroll in another study of an investigational agent prior to completion of Day 42 of the study;
7. Able to take ARAKODA according to Prescribing Information
8. Have been symptomatic no longer than 7 days inclusive of Day 1 when the first dose of study medication is administered.
9. If female, agree to use an acceptable method of birth control from the time of consent through 56 days after the last dose of study drug.
10. Possess a smart phone or tablet, or are willing to utilize a sponsor-provided device if available.

Exclusion Criteria:

1. Have any of the contraindications for ARAKODA in the prescribing information including:

   1. G6PD deficiency
   2. Breastfeeding
   3. Psychotic disorder or current psychotic symptoms
   4. Known hypersensitivity reaction to TQ
2. Evidence of severe or critical illness, defined by at least one of the following:

   1. Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥30 breaths per minute, heart rate ≥125 beats per minute, SpO2 ≤93% on room air
   2. Respiratory failure defined based on resource utilization requiring at least one of the following: i. Endotracheal intubation and mechanical ventilation, oxygen delivered by high flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥0.5), noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO), or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation); ii. Shock (defined by systolic blood pressure <90 mmHg, or diastolic blood pressure <60 mmHg or requiring vasopressors); iii. Multi-organ dysfunction/failure
3. Any other clinically significant acute illness unrelated to COVID-19 within seven days prior to first study drug administration;
4. Receipt of any approved or experimental small molecule treatment for COVID-19 (FDA-approved, off-label, compassionate use, or study-related) within the 30 days prior to the time of the screening evaluation
5. Receipt of any approved or experimental biologic therapeutic for COVID-19 (FDA-approved, off-label, compassionate use, or study-related) within the 90 days prior to the time of the screening evaluation
6. Have been diagnosed (and confirmed by PCR or rapid antigen test) with COVID-19 in the 90 days prior to randomization (other than for this infection);
7. Any excluded concomitant medication as described in the ARAKODA package insert. Receipt of a COVID-19 vaccine is not exclusionary;
8. Any COVID-19 symptoms which, in the opinion of the investigator, is suggestive of possible requirement to hospitalize within 48 hours of enrollment.
9. Positive pregnancy test;
10. Are ≥65 years of age and have a clinical frailty score > 5;
11. Have cystic fibrosis;
12. Have received a transplant;
13. Known to be infected with human immunodeficiency virus (HIV);
14. Have received any B-Cell depleting monoclonal antibody in the last six months;
15. Have a disease or condition which in the opinion of the investigator presents an unacceptable risk of disease progression;
16. Have an aggregate symptom score ≥ 15 and any one of the following risk factors for COVID-19 disease progression: Obesity (BMI ≥31), are a smoker, have never been vaccinated for COVID-19, diabetes with complications, dementia or other neurocognitive disorders, chronic kidney disease, chronic liver disease, COPD or other chronic lung disease, bronchiectasis, coronary atherosclerosis and other heart disease, stroke or other cerebrovascular disease, sickle cell disease or thalassemia, current mood disorder or depression, substance abuse disorder, tuberculosis, cancer that is not invasive squamous and basal carcinomas of the skin or prostate cancer under active surveillance;
17. Have two or more of the following risk factors for COVID-19 disease progression: Obesity (BMI ≥31), are a smoker, diabetes with complications, dementia or other neurocognitive disorders, chronic kidney disease, chronic liver disease, COPD or other chronic lung disease, bronchiectasis, coronary atherosclerosis and other heart disease, stroke or other cerebrovascular disease, sickle cell disease or thalassemia, current mood disorder or depression, substance abuse disorder, tuberculosis, cancer that is not invasive squamous and basal carcinomas of the skin or prostate cancer under active surveillance;
18. Have an aggregate symptom score >32.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-04-27 (Estimated); Study Completion 2024-04-27 (Estimated)

PRIMARY OUTCOMES:
Time to sustained clinical recovery from COVID-19 symptoms (4 uninterrupted days of aggregate symptom scores ≤ 2) through Day 28 (± 2 days) | Day 28 (± 2 days)

SECONDARY OUTCOMES:
MCP-1 levels at Days 5, 14 (± 1 day) and 28 (± 2 days) | Days 5, 14 (± 1 day) and 28 (± 2 days)
Day 5 aggregate symptom score (FDA's 14 COVID-19 symptoms) | Day 5
Time to clinical resolution (uninterrupted daily aggregate symptom score ≤ 2 for at least 1, 2 or 3 occasions) of all COVID-19 symptoms through Day 28 (± 2 days) | Day 28 (± 2 days)
Time to sustained clinical resolution (uninterrupted daily aggregate symptom score ≤ 2 for at least 1, 2, 3, or 4 occasions) of all COVID-19 symptoms through Days 14 (± 1 day) and 42 (± 2 days) | Days 14 (± 1 day) and 42 (± 2 days)
Proportion of patients with sustained clinical resolution (uninterrupted daily aggregate symptom score ≤ 2 on at least 1, 2, or 3 or 4 occasions) of all COVID-19 symptoms at Days 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days) | Days 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days)
Time to first instance of clinical recovery from fever, cough, and shortness of breath at 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days) who reported at least one such symptom on Day 1 (recovery defined as in Dow and Smith 2022) | 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days)
Proportion of patients recovered (first instance) from cough, fever, and shortness of breath at Day 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days) who reported at least one such symptom on Day 1 (recovery defined as in Dow and Smith 2022) | Day 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days)
Time to sustained recovery (two, three or four uninterrupted days of recovery) from fever, cough, and shortness of breath at 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days) who reported at least one such symptom on Day 1 | 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days)
Proportion of patients recovered (sustained recovery for two, three or four uninterrupted days) from cough, fever, and shortness of breath at Day 14 (± 1 day), Day 28 (± 1 day) and 42 (± 2 days) who reported at least one such symptom on Day 1 | Day 14 (± 1 day), Day 28 (± 1 day) and 42 (± 2 days)

OTHER OUTCOMES:
Proportion of patients with negative COVID-19 rapid antigen test at Day 7 (± 1 day) and at first report after day 3 of feeling able to resume normal activities (± 1 days) | Day 7 (± 1 day) and at first report after day 3 of feeling able to resume normal activities (± 1 days)
Clinical relapse through Day 42 (± 2 days) of COVID symptoms defined as at least three days of aggregate symptoms score > 2 after achieving clinical recovery for the primary endpoint | Day 42 (± 2 days)
Time to first report by the patient that they can resume normal activities | Time to first report by the patient
Time to first report by the patient that they feel recovered from COVID-19 symptoms | Time to first report by the patient
Cytokine and chemokine levels at Screening, Day 5, Day 14 (± 1 day) and Day 28 (± 2 days) | Screening, Day 5, Day 14 (± 1 day) and Day 28 (± 2 days)
Total anti-SARS-CoV-2 spike protein antibody levels (IgM and IgG) at Screening and Day 14 (± 1 day) | Screening and Day 14 (± 1 day)
Hospitalization rates due to COVID-19 symptoms (excluding non-COVID 19 causes including admittance for other upper respiratory infections and admittance only for administrative or observations purposes) | Day 42 (± 2 days)
Number of unscheduled COVID-19-related medical visits (Doctor's office or emergency room (ER) visit) | Day 42 (± 2 days)
Incidence of COVID-19 related neuropsychiatric symptoms (depression, anxiety, impaired wakefulness, memory or ability thinking) | Incidence of COVID-19 related neuropsychiatric symptoms
Time to first instance of and sustained recovery from "Long Covid" symptoms individually and together | Time to first instance of and sustained recovery
Proportion of patients recovered from "Long Covid" symptoms individually and together at Days 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days) | Days 14 (± 1 day), 28 (± 2 days) and 42 (± 2 days)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 60º Pharmaceuticals LLC. Clinical Study Report, TQ 2020_06. A double-blind placebo-controlled study to assess the efficacy and safety of oral tafenoquine versus placebo in patients with mild to moderate COVID-19 disease. 14 July 2022
- [Result] Bobrowski T, Chen L, Eastman RT, Itkin Z, Shinn P, Chen CZ, Guo H, Zheng W, Michael S, Simeonov A, Hall MD, Zakharov AV, Muratov EN. Synergistic and Antagonistic Drug Combinations against SARS-CoV-2. Mol Ther. 2021 Feb 3;29(2):873-885. doi: 10.1016/j.ymthe.2020.12.016. Epub 2020 Dec 15. PMID 33333292
- [Result] Brueckner RP, Lasseter KC, Lin ET, Schuster BG. First-time-in-humans safety and pharmacokinetics of WR 238605, a new antimalarial. Am J Trop Med Hyg. 1998 May;58(5):645-9. doi: 10.4269/ajtmh.1998.58.645. PMID 9598455
- [Result] Chen Y, Yang WH, Chen HF, Huang LM, Gao JY, Lin CW, Wang YC, Yang CS, Liu YL, Hou MH, Tsai CL, Chou YZ, Huang BY, Hung CF, Hung YL, Wang WJ, Su WC, Kumar V, Wu YC, Chao SW, Chang CS, Chen JS, Chiang YP, Cho DY, Jeng LB, Tsai CH, Hung MC. Tafenoquine and its derivatives as inhibitors for the severe acute respiratory syndrome coronavirus 2. J Biol Chem. 2022 Mar;298(3):101658. doi: 10.1016/j.jbc.2022.101658. Epub 2022 Jan 29. PMID 35101449
- [Result] Dow GS, Luttick A, Fenner J, Wesche D, Yeo KR, Rayner C. Tafenoquine inhibits replication of SARS-CoV-2 at pharmacologically relevant cincentrations in vitro. Biorxiv; Tafenoquine inhibits replication of SARS-Cov-2 at pharmacologically relevant concentrations in vitro. bioRxiv.2020. https://doi.org/10.1101/2020.07.12.199059
- [Result] Dow GS, Smith BL. A phase II, double blind, placebo-controlled, randomized evaluation of the safety and efficacy of tafenoquine in patients with mild-moderate COVID-19 disease. New Microbes New Infect. 2022 Jun 1;47:100986. doi: 10.1016/j.nmni.2022.100986. eCollection 2022 Apr-May. PMID 35668841
- [Result] Grassin-Delyle S, Salvator H, Brollo M, Catherinot E, Sage E, Couderc LJ, Naline E, Devillier P. Chloroquine Inhibits the Release of Inflammatory Cytokines by Human Lung Explants. Clin Infect Dis. 2020 Nov 19;71(16):2265-2268. doi: 10.1093/cid/ciaa546. PMID 32382733
- [Result] Sato R, Imaizumi T, Aizawa T, Watanabe S, Tsugawa K, Kawaguchi S, Seya K, Matsumiya T, Tanaka H. Inhibitory effect of anti-malarial agents on the expression of proinflammatory chemokines via Toll-like receptor 3 signaling in human glomerular endothelial cells. Ren Fail. 2021 Dec;43(1):643-650. doi: 10.1080/0886022X.2021.1908901. PMID 33820486
- [Result] Shivakumar S, Panigrahi T, Shetty R, Subramani M, Ghosh A, Jeyabalan N. Chloroquine Protects Human Corneal Epithelial Cells from Desiccation Stress Induced Inflammation without Altering the Autophagy Flux. Biomed Res Int. 2018 Nov 1;2018:7627329. doi: 10.1155/2018/7627329. eCollection 2018. PMID 30519584
- [Result] Song Y, Zhang H, Zhu Y, Zhao X, Lei Y, Zhou W, Yu J, Dong X, Wang X, Du M, Yan H. Lysozyme Protects Against Severe Acute Respiratory Syndrome Coronavirus 2 Infection and Inflammation in Human Corneal Epithelial Cells. Invest Ophthalmol Vis Sci. 2022 Jun 1;63(6):16. doi: 10.1167/iovs.63.6.16. PMID 35713893
- [Result] United States Centers for Disease Control. Daily update of COVID-19 cases. Accessed on 19 February 2023 at https://covid.cdc.gov/covid-data-tracker/#datatracker-home.